CLINICAL TRIAL: NCT05346081
Title: Pulmonary Function Assessment and Evaluation Using Self-administrable and Portable Electrical Impedance Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok Wang Chun, Resident Speicalist, Queen Mary Hospital, Hong Kong
Other Study IDs: UW 21-644
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with underlying lung disease
  Interventions: Device: Electrical impedance tomography
- Healthy subjects
  Interventions: Device: Electrical impedance tomography

INTERVENTIONS:
Device: Electrical impedance tomography — Electrical impedance tomography (EIT) is a potential alternative non-invasive diagnostic screening measure to spirometry.

SUMMARY:
Spirometry is the most commonly used modality for measuring lung function. However, spirometry is a coordination-dependent test and may lead to erroneous results if subjects are unable to fully comply with the instructions. It also lacks the capability for regional assessment of pulmonary functions.

Electrical impedance tomography (EIT) is a potential alternative test to spirometry. EIT has been employed in clinical use to provide qualitative and quantitative measurements of ventilation in patients on mechanical ventilators to prevent lung damage or patient-ventilator desynchronies.

In this study, we aim to utilize EIT lung device to study EIT-derived indicators in pulmonary functional assessment and develop novel biomarkers for detecting and monitoring pulmonary diseases. This is a non-interventional clinical study on patients with chronic lung diseases, to establish the feasibility of using EIT-lung device in detecting lung functional changes. Specifically, we will establish the relationship between EIT-derived functional indicators and spirometry results. Furthermore, we will explore, develop, and establish EIT-derived regional lung functional indicators in healthy and chronic diseased states.

Subjects with underlying lung disease, and age- and gender-matched healthy control subjects will be recruited in this study. They will perform spirometry and EIT examination, as well as an interview with a structured questionnaire.

The results from spirometry and EIT test will be correlated and compared to identify the feasibility and accuracy of EIT lung device. Lung function parameters (e.g. FEV1, FVC, and FEV1/FVC ratio) measured using a spirometer would also be calculated from lung flow-volume curves derived from continuous EIT functional images. Regional lung function assessment will also be explored using EIT, and establish regional EIT features that could assist in screening and evaluating different chronic lung diseases. The EIT-derived indicators will be finally analyzed together with demographics, clinical assessments and patient history to derive fine grained insights and elucidate the effect of demographics and biometrics on EIT lung data. The parameters include, but not limited to, age, chest size, gender, weight, height, BMI, smoking habits and ethnicity. The analysis will improve the stability of the EIT indicators, and ultimately increase their predictive power towards diseased lung regions.

With the availability of the EIT device on lung function assessment, which was validated with spirometry findings, patients who are unable to perform spirometry but need a proper lung function assessment can benefit by having the EIT test. These patients include but not limited to those who need major lung resection and interstitial lung diseases on anti-fibrotic. EIT can also be a more comfortable alternative to spirometry for patients who need lung function assessment.

ELIGIBILITY:
Inclusion Criteria:

Pulmonary disease subjects Patients of age 18 to 75 suspected or diagnosed with pulmonary diseases scheduled to undergo standard pulmonary function test will be recruited. These patients will undergo an interview (with a structured questionnaire), Pulmonary Functional Test (PFT) and EIT examination.

Healthy control subjects Healthy adults of age 18 to 75 who do not have any known pulmonary diseases will be examined. These healthy individuals will undergo spirometry and EIT examination, as well as an interview with a structured questionnaire to ensure they do not have any clinical features or symptoms.

Exclusion Criteria:

* Subjects with implanted electronic devices, in case EIT might interfere with the devices
* Subjects with spinal diseases
* Subjects with unstable cardiac or respiratory conditions
* Pregnant women
* Patients who are unable to perform spirometry

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Pulmonary disease subjects Patients of age 18 to 75 suspected or diagnosed with pulmonary diseases scheduled to undergo standard pulmonary function test will be recruited. These patients will undergo an interview (with a structured questionnaire), Pulmonary Functional Test (PFT) and EIT examination.
  Healthy control subjects Healthy adults of age 18 to 75 who do not have any known pulmonary diseases will be examined. These healthy individuals will undergo spirometry and EIT examination, as well as an interview with a structured questionnaire to ensure they do not have any clinical features or symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional test comparison between spirometry and EIT lung device: | 31/12/2022
  This study will elucidate the feasibility of EIT in testing lung function in patients and compare its outcomes with the spirometry tests. We expect that the global EIT-derived functional parameters corroborate with spirometry results.
Regional lung function assessment in patients | 31/12/2022
  Regional EIT-derived structural and functional biomarkers of patients and healthy controls will be analyzed. This will potentially establish EIT-derived biomarkers for different chronic lung diseases.
Effect of demographics, clinical assessments and patient history on EIT measurements | 31/12/2022
  EIT derived indicators will be finally analyzed together with demographics, clinical assessments (including CT scans if available) and patient history to derive fine grained insights for potential early detection and treatment monitoring of different chronic lung diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided